CLINICAL TRIAL: NCT03123055
Title: A Multi-Center, Open-Label Phase 1b/2 Study of a Novel FGFR3 Inhibitor (B-701) Combined With Pembrolizumab in Subjects With Locally Advanced or Metastatic Urothelial Carcinoma Who Have Progressed Following Platinum-based Chemotherapy
Brief Title: A Study of B-701 in Combination With Pembrolizumab in Treatment of Locally Advanced or Metastatic Urothelial Cell Carcinoma
Acronym: FIERCE-22
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: program has been put on hold by the sponsor
Sponsor: Rainier Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B-701-U22; 2017-001292-23 (EudraCT Number)
Record Dates: First submitted 2017-04-11; First posted 2017-04-21 (Actual); Results first posted 2020-03-18 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2020-02

CONDITIONS: Locally Advanced or Metastatic Urothelial Cell Carcinoma; Urinary Bladder Disease; Urological Diseases
Keywords: Urothelial Cell Carcinoma; UCC; bladder cancer; B-701; FGFR3; invasive bladder cancer; Transitional Cell Carcinoma; TCC; second line therapy; monoclonal antibody; combination therapy; Phase 1b; pembrolizumab; checkpoint inhibitor; Phase 2; Urothelial Carcinoma; Vofatamab
MeSH Terms: conditions — Urinary Bladder Diseases; Urologic Diseases; Urinary Bladder Neoplasms; Carcinoma, Transitional Cell | interventions — B701 protein, Human herpesvirus 6; vofatamab; pembrolizumab

STUDY DESIGN:
Intervention Model Description: B-701 (vofatamab) as monotherapy for first 2 weeks followed by B-701 (vofatamab) in combination with pembrolizumab thereafter.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- B-701 (vofatamab) (Experimental): B-701 (vofatamab, 25 mg/kg) will be administered via IV infusion on Cycle 0 Day 1 for a single 14-day cycle.
  Interventions: Drug: B-701
- B-701 (vofatamab) plus pembrolizumab (Experimental): B-701 (vofatamab, 25 mg/kg [or the recommended Phase 2 dose if different than 25 mg/kg]) plus pembrolizumab (200 mg) will be administered by IV infusion on Cycle 1 Day 1 once every 3 weeks.
  Interventions: Drug: B-701; Drug: Pembrolizumab

INTERVENTIONS:
Drug: B-701 — B-701 (vofatamab) is a human IgG1 monoclonal antibody that is highly specific for the FGFR3 receptor.
  Other Names: MFGR1877S; Vofatamab
Drug: Pembrolizumab — Pembrolizumab is a humanized antibody used in cancer immunotherapy. Pembrolizumab targets and blocks a protein called PD-1 on the surface of certain immune cells called T-cells. Blocking PD-1 triggers the T-cells to find and kill cancer cells.
  Other Names: Keytruda
  Arms: B-701 (vofatamab) plus pembrolizumab

SUMMARY:
This is a Phase 1b/2 multi-center, open-label study to establish the initial safety and to determine a recommended Phase 2 dose of B-701 in combination with pembrolizumab, and to determine safety, tolerability and efficacy of B-701 (vofatamab) plus pembrolizumab in the treatment of subjects with locally advanced or metastatic UCC, who have progressed following platinum-based chemotherapy and who have not received prior immune checkpoint inhibitor therapy.

DETAILED DESCRIPTION:
This is a Phase 1b/2 multi-center, open-label study to determine the safety, tolerability, and efficacy of B-701 (vofatamab) plus pembrolizumab in the treatment of subjects with locally advanced or metastatic UCC, who have progressed following platinum-based chemotherapy and who have not received prior immune checkpoint inhibitor or FGFR inhibitor-targeted therapy. The study consists of 2 parts: a Phase 1b lead-in phase enrolling 6 to 18 subjects and a Phase 2 dose expansion phase enrolling up to a total of 74 subjects.

Subjects who discontinue B-701 (vofatamab) may continue on study and receive pembrolizumab alone until disease progression, death, withdrawal of patient consent, or study termination. Subjects who discontinue pembrolizumab may continue on study and receive B-701 (vofatamab) alone until disease progression, death, withdrawal of patient consent, or study termination.

ELIGIBILITY:
Key Inclusion Criteria:

1. Have locally advanced (on TNM staging: T4b and any N, or any T and N2-3) or metastatic transitional cell carcinoma of the urothelium, including of the urinary bladder, urethra, ureter, and/or renal pelvis. The diagnosis must be histologically or cytologically confirmed.
2. Have progression during or following platinum-containing chemotherapy or within 12 months of neoadjuvant or adjuvant treatment with platinum-containing chemotherapy.
3. Have available archival tumor or be willing to undergo diagnostic biopsy at screening. Sample must be of suitable quality and quantity to satisfy group assignment and biomarker endpoints.
4. Have measurable disease according to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1).
5. Eastern Cooperative Oncology Group (ECOG) performance status (PS) ≤ 1.

Key Exclusion Criteria:

1. Participants with a history of idiopathic pulmonary fibrosis, organizing pneumonia, drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis on the Screening chest CT scan.
2. Prior therapy with an anti-programmed cell death 1 (PD-1) or anti-PD-Ligand 1 agent, or with an agent directed to another co-inhibitory T-cell receptor or FGFR inhibitor.
3. Patients with autoimmune disease or medical conditions that required systemic corticosteroids (> 10 mg/day prednisone or its equivalent) or other immunosuppressive medications or any other form of systemic immunosuppressive therapy within 7 days prior to the first dose of study treatment. Note: Replacement therapy (e.g. physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
4. Primary central nervous system (CNS) malignancy or CNS metastases.
5. History of clinically significant coagulation or platelet disorder in the past 12 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2017-04-20 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rainier Therapeutics, Study Chair — Rainier Therapeutics
Locations (46):
- United States (8):
  - Research Site, Greenbrae, California
  - Research Site, Fort Wayne, Indiana
  - Research Site, Louisville, Kentucky
  - Washington University School of Medicine, St Louis, Missouri
  - Research Site, Cleveland, Ohio
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Germantown, Tennessee
  - Research Site, Houston, Texas
- Belgium (3):
  - Research Site, Brussels
  - Research Site, Leuven
  - Research Team, Yvoir
- Research Team, Copenhagen, Denmark
- France (2):
  - Research Site, Bordeaux
  - Research Site, Dijon
- Germany (6):
  - Research Site, Dresden
  - Research Site, Frankfurt
  - Research Site, Heidelberg
  - Research Site, Kassel
  - Research Site, Munich
  - Research Site, Münster
- Research Site, Budapest, Hungary
- Research Site, Milan, Italy
- Research Site, Chisinau, Moldova
- Research Site, Utrecht, Netherlands
- Poland (4):
  - Research Site, Katowice
  - Research Site, Warsaw
  - Research Site, Wieliszew
  - Research Site, Wroclaw
- Russia (3):
  - Research Site, Moscow
  - Research Site, Saint Petersburg
  - Research Team, Ufa
- Serbia (4):
  - Research Site, Belgrade
  - Research Site, Kamenitz
  - Research Site, Kragujevac
  - Research Site, Niš
- South Korea (3):
  - Research Site, Gwangju
  - Research Site, Seongnam-si
  - Research Site, Seoul
- Spain (3):
  - Research Site, Madrid, CA
  - Research Site, Barcelona
  - Research Site, Madrid
- Research Site, Uppsala, Sweden
- Turkey (Türkiye) (2):
  - Research Site, Ankara
  - Research Site, Antalya
- Ukraine (2):
  - Research Site, Dnipro
  - Research Site, Kyiv

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase 2: B-701 (vofatamab, 25 mg/kg plus pembrolizumab (200 mg) will be administered by IV infusion on Cycle 1 Day 1 once every 3 weeks.
Period: Overall Study
Arm/Group | Phase 2
Started | 28
Completed | 28
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Phase 2
Number analyzed (Participants) | 28
Age, Continuous [Median (Full Range); unit: years] | 61.5 [21 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 27
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities Within a Period of 35 Days
Description: Number of Participants with Dose Limiting Toxicities within a period of 35 days will be analyzed reviewing the aggregate of adverse events (AEs) and serious adverse events (SAEs) by the B-701 program Safety Oversight Committee and will result in a recommended Phase 2 dose. Six subjects at a time are enrolled and observed for 35 days after the initial dose. If 2 or more subjects experience a DLT that dose will be declared intolerable and de-escalation of the dose will occur.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Groups:
- B-701 (Vofatamab) Plus Pembrolizumab: B-701 (vofatamab) plus pembrolizumab (200 mg) will be administered by IV infusion on Cycle 1 Day 1 once every 3 weeks in a 6+6 dose escalation designed to determine the RP2D of the combination.
Arm/Group | B-701 (Vofatamab) Plus Pembrolizumab
Number analyzed (Participants) | 8
Participants | 0

2. Primary Outcome: Number of Subjects Experiencing Adverse Events (AEs and SAEs)
Description: Evaluate the safety and tolerability of B-701 (vofatamab) plus pembrolizumab in subjects with UCC as assessed by number of subjects experiencing adverse events (AEs and SAEs), physical examination findings, laboratory test results, and vital signs over time. This outcome is measured by a safety monitoring committee who regularly met and reviewed aggregate trends of reports AEs, lab ranges, physical exams etc. and determined if the drug was safe to continue.
Time Frame: 2.5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2
Number analyzed (Participants) | 28
Participants | 28

3. Primary Outcome: Efficacy of B-701 (Vofatamab) Plus Pembrolizumab Measured by ORR
Description: Evaluate the efficacy of B-701 (vofatamab) plus pembrolizumab in subjects with UCC as measured by objective response rate (ORR) by RECIST 1.1. ORR is defined as the percentage of subjects who have baseline measurable disease and who achieve a best response of either complete response (CR) or partial response (PR).
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2
Number analyzed (Participants) | 22
Participants | 9

4. Secondary Outcome: Assessment of Changes in Biomarkers Induced by B-701 (Vofatamab)
Description: Whole blood (PBMCs), serum, and plasma samples for biomarker analyses will be obtained prior to infusion of B-701 at pre-defined visit days.
  The effects of B-701 on the downstream signaling of the FGFR3 pathway, tumor sub-type and on the immune surveillance of UCC tumors will be monitored using techniques that include gene expression profiling (such as whole transcriptome RNAseq), sequencing of T-cell receptors, and immunohistochemistry.
Time Frame: 2.5 years
Population: The study was terminated early and this outcome was not analyzed because the data were not collected.
Arm/Group | Phase 2
Number analyzed (Participants) | 0

5. Secondary Outcome: Efficacy of B-701 (Vofatamab) in Combination With Pembrolizumab as Measured by DOR
Description: Evaluate the efficacy of B-701 (vofatamab) in combination with pembrolizumab in the treatment of subjects with UCC as measured by duration of objective response (DOR), defined as the time from first occurrence of a documented, objective response until the time of relapse or death from any cause (RECIST 1.1).
Time Frame: 2 years
Population: The study was terminated early and this outcome was not analyzed because the data were not collected.
Arm/Group | Phase 2
Number analyzed (Participants) | 0

6. Secondary Outcome: Efficacy of B-701 (Vofatamab) in Combination With Pembrolizumab as Measured by DCR
Description: Evaluate the efficacy of B-701 in combination with pembrolizumab in the treatment of subjects with UCC as measured by disease control rate (DCR), defined as the percentage of subjects who achieve either complete response (CR) or partial response (PR) or stable disease (SD) according to RECIST 1.1.
Time Frame: 2 years
Population: The study was terminated early and this outcome was not analyzed because the data were not collected.
Arm/Group | Phase 2
Number analyzed (Participants) | 0

7. Secondary Outcome: Efficacy of B-701 (Vofatamab) in Combination With Pembrolizumab as Measured by PFS
Description: Evaluate the efficacy of B-701 (vofatamab) in combination with pembrolizumab in the treatment of subjects with UCC as measured by progression-free survival (PFS), defined as the time from a first study treatment dose to first occurrence of disease progression (per RECIST 1.1) or death from any cause, whichever occurs first.
Time Frame: 2 years
Population: The study was terminated early and this outcome was not analyzed because the data were not collected.
Arm/Group | Phase 2
Number analyzed (Participants) | 0

8. Secondary Outcome: Efficacy of B-701 (Vofatamab) in Combination With Pembrolizumab as Measured by OS
Description: Evaluate the efficacy of B-701 (vofatamab) in combination with pembrolizumab in the treatment of subjects with UCC as measured by overall survival (OS), defined as the time from first study drug administration to death from any cause (RECIST 1.1)
Time Frame: 2.5 years
Population: The study was terminated early and this outcome was not analyzed because the data were not collected.
Arm/Group | Phase 2
Number analyzed (Participants) | 0

9. Secondary Outcome: Change in Subject Reported Quality of Life
Description: Evaluate the efficacy of B-701 (vofatamab) in combination with pembrolizumab in the treatment of subjects with UCC as measured by the change over time in subject reported quality of life as measured by the European Organization for Research and Treatment Quality of Life Questionnaire (EORTC QLQ-C30).
Time Frame: 2 years
Population: The study was terminated early and this outcome was not analyzed because the data were not collected.
Arm/Group | Phase 2
Number analyzed (Participants) | 0

10. Other Pre Specified Outcome: PK Analysis of B-701 (Vofatamab)
Description: PK will be analyzed by measuring B-701 C(trough) levels. B-701 C(trough) levels then will be summarized over time throughout the study and will be compared to predicted B-701 C(trough) levels, whose prediction is based on data observed in previous studies with B-701.
Time Frame: 2 years
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Immunogenicity of B-701 (Vofatamab)
Description: Determine the immunogenicity of B-701 as measured by anti-B-701 antibody titers at several time points throughout the study.
Time Frame: 2 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of consent through 30 days after the last dose of study drug.
Arm/Group | Phase 2
All-Cause Mortality (participants affected / at risk) | 12/28
Serious Adverse Events (participants affected / at risk) | 13/28
Other Adverse Events (participants affected / at risk) | 28/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 2 (N=28)
Pyrexia (General disorders) | 1 (1)
Sudden death (General disorders) | 1 (1)
Bacteraemia (Infections and infestations) | 1 (1)
Gastroenteritis Escherichia coli (Infections and infestations) | 1 (1)
Kidney Infection (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 2 (2)
Tracheobronchitis (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2)
Urosepsis (Infections and infestations) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1)
Paraneoplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Embolism (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 2 (N=28)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Acute on chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Acute renal insufficiency (Renal and urinary disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
ALP increased (Investigations) | 1 (1)
ALT increased (Investigations) | 3 (3)
Anemia (Blood and lymphatic system disorders) | 7 (7)
Anemia aggravated (Blood and lymphatic system disorders) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Appetite lost (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
AST increased (Investigations) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Basilar atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bladder infection (Infections and infestations) | 1 (1)
Bladder pain (Renal and urinary disorders) | 1 (1)
Bloody vaginal discharge (Reproductive system and breast disorders) | 1 (1)
Breast nodule (Reproductive system and breast disorders) | 1 (1)
Breast pain (Reproductive system and breast disorders) | 1 (1)
Burning esophagus (Gastrointestinal disorders) | 1 (1)
Burning in eyes (Eye disorders) | 1 (1)
Cachexia (Metabolism and nutrition disorders) | 1 (1)
Cataracts (Eye disorders) | 1 (1)
Chills (General disorders) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 1 (1)
Common cold (Infections and infestations) | 2 (2)
Confusion (Psychiatric disorders) | 1 (1)
Congestive heart failure (Cardiac disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Crackles lung (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cramps in legs (Musculoskeletal and connective tissue disorders) | 1 (1)
C-reactive protein increased (Investigations) | 1 (1)
Creatinine increased (Investigations) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 6 (6)
Dizziness aggravated (Nervous system disorders) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea exacerbated (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1)
Edema limbs (General disorders) | 1 (1)
Elevated liver enzymes (Investigations) | 1 (1)
Erythema facial (Skin and subcutaneous tissue disorders) | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 1 (1)
Fatigue (General disorders) | 7 (7)
Fatigue aggravated (General disorders) | 1 (1)
Fever (General disorders) | 4 (4)
Flushing (Vascular disorders) | 1 (1)
Forgetfulness (Nervous system disorders) | 1 (1)
General body pain (General disorders) | 1 (1)
General physical health deterioration (General disorders) | 1 (1)
Glucose intolerance (Metabolism and nutrition disorders) | 1 (1)
Gonalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 2 (2)
Hunger (General disorders) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2)
Hypertension arterial (Vascular disorders) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 1 (1)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Itching eyes (Eye disorders) | 1 (1)
Kidney failure (Renal and urinary disorders) | 2 (2)
Kidney infection (Infections and infestations) | 1 (1)
Kidney pain (Renal and urinary disorders) | 1 (1)
Knee arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Lateral myocardial infarction (Cardiac disorders) | 1 (1)
Leg edema (General disorders) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1)
Loose stools (Gastrointestinal disorders) | 1 (1)
Lower abdominal pain (Gastrointestinal disorders) | 1 (1)
Lumbar pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Lymphadenitis (Blood and lymphatic system disorders) | 1 (1)
Muscle cramps (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia of lower extremities (Musculoskeletal and connective tissue disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 3 (3)
Nausea aggravated (Gastrointestinal disorders) | 1 (1)
NT-proBNP increased (Investigations) | 1 (1)
Ophthalmic migraine (Nervous system disorders) | 1 (1)
Oral candidiasis (Infections and infestations) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in foot (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in lumbar spine (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain pelvic (Reproductive system and breast disorders) | 1 (1)
Painful R arm (Musculoskeletal and connective tissue disorders) | 1 (1)
Paresthesia lower limb (Nervous system disorders) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 1 (1)
Phlegmon (Infections and infestations) | 1 (1)
Platelet count low (Investigations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Procalcitonin increased (Investigations) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1)
Rash all over (Skin and subcutaneous tissue disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2)
Renal calculi (Renal and urinary disorders) | 1 (1)
Respiratory tract infection viral (Infections and infestations) | 1 (1)
Restless leg syndrome (Nervous system disorders) | 1 (1)
Shoulder blade pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Shoulder pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Skin burning sensation (Skin and subcutaneous tissue disorders) | 1 (1)
Skin rash (Skin and subcutaneous tissue disorders) | 2 (2)
Skin red (Skin and subcutaneous tissue disorders) | 1 (1)
Slurred speech (Nervous system disorders) | 1 (1)
Stomach pain (Gastrointestinal disorders) | 1 (1)
Streptococcal infection (Infections and infestations) | 1 (1)
Subfebrile (General disorders) | 1 (1)
Swallowing difficult (Gastrointestinal disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Taste changed (Nervous system disorders) | 1 (1)
Thirst (General disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Tongue black (Gastrointestinal disorders) | 1 (1)
Tremor of hands (Nervous system disorders) | 1 (1)
Troponin increased (Investigations) | 1 (1)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Type I diabetes mellitus (Metabolism and nutrition disorders) | 1 (1)
Unilateral leg pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Upper abdominal tenderness (Gastrointestinal disorders) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Ureterohydronephrosis (Renal and urinary disorders) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 2 (2)
Urinary tract infection (Infections and infestations) | 1 (1)
Urinary urgency (Renal and urinary disorders) | 1 (1)
Urination pain (Renal and urinary disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2)
WBC increased (Investigations) | 1 (1)
Weakness (General disorders) | 1 (1)
Weakness worsened (General disorders) | 1 (1)
Weight loss (Investigations) | 3 (3)
Weight loss poor (Metabolism and nutrition disorders) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-01): https://cdn.clinicaltrials.gov/large-docs/55/NCT03123055/Prot_SAP_000.pdf